CLINICAL TRIAL: NCT00004364
Title: Study of Novel Types of Familial Diabetes Insipidus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11939; NU-570
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Diabetes Insipidus
Keywords: diabetes insipidus; endocrine disorders; rare disease
MeSH Terms: conditions — Diabetes Insipidus; Endocrine System Diseases; Rare Diseases | interventions — Deamino Arginine Vasopressin

INTERVENTIONS:
Drug: desmopressin

SUMMARY:
OBJECTIVES:

I. Define the phenotype and genotype of previously unrecognized types of familial diabetes insipidus (FDI) in kindreds with atypical or novel forms of FDI.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Participants undergo a series of tests to determine the presence, absence, cause, natural history, clinical status, and mode of inheritance of their type of diabetes insipidus (DI). The studies include measurements of basal fluid intake and urine output, plasma vasopressin during standard fluid deprivation or waterload/saline infusion tests, and changes in water balance during a therapeutic trial of DDAVP. If clinically indicated, echocardiograms and assays of plasma catecholes and renin are also completed.

Linkage analysis is performed for all participants; kindreds with the Marfan-like syndrome are also studied for the fibrillin-1 genotype.

Participants determined to have DI are treated with desmopressin for 2 days.

ELIGIBILITY:
* Familial diabetes insipidus (DI) in atypical or novel form, e.g.: Dipsogenic DI Neurohypophyseal DI
* Affected and unaffected members of kindreds eligible

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 1995-12

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Robertson, Study Chair — Northwestern University